CLINICAL TRIAL: NCT05281029
Title: A Multicenter, Single-arm, Prospective Observational Study to Evaluate the Safety and Effectiveness of Gemigliptin (as Monotherapy or as Single Pill Combinations) in Patients Aged ≥ 65 Years With Type 2 Diabetes Mellitus
Brief Title: Observational Study Gemigliptin in Patients Aged ≥ 65 Years With Type 2 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Other Study IDs: LG-DPOS002
Record Dates: First submitted 2022-03-06; First posted 2022-03-15 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate safety and effectiveness of treatment with gemigliptin for 24 weeks in Korean patients aged ≥ 65 years with type 2 diabetes mellitus in routine clinical settings

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been started on gemigliptin in accordance with the approved label and who have signed on the consent form

Exclusion Criteria:

* Patients with previous exposure to gemigliptin and current participation in clinical trials

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Primary care clinic, secondary and tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of HbA1c at 24 weeks | Baseline, 24 weeks

SECONDARY OUTCOMES:
Change from Baseline of HbA1c at 12 weeks | Baseline, 12 weeks
The rate of subjects who reached the target value of less than 7% (reasonable HbA1c goal) of HbA1c. | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea